CLINICAL TRIAL: NCT03132337
Title: Biomarkers of Endothelial Dysfunction in Pediatric Patients Receiving High Intensity Chemotherapy/Irradiation
Brief Title: Sinusoidal Obstruction Syndrome for Stem Cell Transplant Patients Biomarker Study
Acronym: SOSBiomarker
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Sophie Paczesny, Professor, Department of Pediatrics, Indiana University
Other Study IDs: 1701020549
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Sinusoidal Obstruction Syndrome
MeSH Terms: conditions — Hepatic Veno-Occlusive Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stem Cell Transplant: Serial Blood Draws
  Interventions: Other: Serial Blood Draws

INTERVENTIONS:
Other: Serial Blood Draws — Day 0 and Day 3 blood draw for SOS biomarkers. If subject develops SOS blood draw prior to dose of Defibrotide, Day 14 after Defibrotide and Day 21 after Defibrotide.

SUMMARY:
The goal of this is to learn more about stem cell transplant and complications that some people have after their transplants, in particular sinusoidal obstruction syndrome (SOS), also called veno-occlusive disease of the liver.

DETAILED DESCRIPTION:
This is a multicenter, prospective, observational trial. We will measure biomarkers and determine thresholds that will predict increased risk for SOS in pediatric patients receiving HCT or high intensity chemotherapy/irradiation with the future goal of a randomized, interventional, open-label, multicenter trial that will test the preemptive use of defibrotide for prevention of SOS in an enriched high-risk population.

ELIGIBILITY:
Inclusion Criteria:

Age ≤ 25 years undergoing HCT for any reason who fulfill any ONE (1) of the following criteria:

1. History of hepatic disease as defined by:

   1. Viral hepatitis (i.e., hepatitis C virus [HCV])
   2. Liver tumor before HCT
   3. Hepatic fibrosis or cirrhosis before HCT as proven by liver biopsy
   4. High aspartate aminotransferase (AST) (> 2x ULN) before HCT (pre-transplant evaluation)
   5. High alanine transaminase (ALT) (> 2x ULN) before HCT
   6. High bilirubin (> 1.2x ULN) before HCT
2. HCT high-risk features including:

   a. Conditioning with high-risk modalities including: i. Busulfan (BU)-containing regimen particularly with oral BU + cyclophosphamide ii. TBI-containing regimen, particularly cyclophosphamide + total-body irradiation (TBI) b. ≥ 2 HCT c. Allo-HCT for leukemia > or = second relapse d. Unrelated donor (URD) HCT e. Human leukocyte antigen (HLA) mismatch HCT (less than 10 of 10 for bone marrow/peripheral blood stem cell [BM/PBSC] or anything less than 6 of 6 for UCB) f. Use of sirolimus + tacrolimus prophylaxis for GVHD
3. High-risk disease states including:

   1. Juvenile myelo-monocytic chronic leukemia (JMML)
   2. Primary hemophagocytic lymphohistiocytosis (HLH)
   3. Adrenoleukodystrophy
   4. Osteopetrosis
4. Other high-risk features including:

   1. Prior treatment with gemtuzumab ozogamicin
   2. Use of hepatotoxic drugs 1 month before HCT and during HCT
   3. Iron overload (i.e., thalassemia/sickle cell) with serum ferritin > 1000ng/ml
   4. Deficit of ATIII, T-PA (i.e., < 30% normal values), and resistance to activated protein C if clinical indication (these values do not have to be specifically checked if no clinical history)
   5. Young age < 2 years but more than 1 month

Exclusion Criteria:

Patients who are transplanted but do not fulfill any of the above mentioned criteria.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Stem Cell Transplant patients
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
SOS proteomic markers | Until the end of the study evaluation, day 180
  Measure for 3 SOS proteomic markers, L-Ficolin, HA, and ST2, as early predictors of SOS incidence through study completion.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Indiana University, Indianapolis, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Han Y, Bidgoli A, DePriest BP, Mendez A, Bijangi-Vishehsaraei K, Perez-Albuerne ED, Krance RA, Renbarger J, Skiles JL, Choi SW, Liu H, Paczesny S. Prospective assessment of risk biomarkers of sinusoidal obstruction syndrome after hematopoietic cell transplantation. JCI Insight. 2023 May 22;8(10):e168221. doi: 10.1172/jci.insight.168221. PMID 37071469